CLINICAL TRIAL: NCT03712228
Title: A Multicenter, Randomized, Placebo-controlled, Parallel-arm Study to Investigate the Efficacy, Pharmacokinetics, and Safety of CSL312 in Subjects With Hereditary Angioedema
Brief Title: A Study to Investigate CSL312 in Subjects With Hereditary Angioedema (HAE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CSL312_2001; 2018-000605-24 (EudraCT Number)
Record Dates: First submitted 2018-10-17; First posted 2018-10-19 (Actual); Results first posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Hereditary Angioedema
MeSH Terms: conditions — Angioedemas, Hereditary

STUDY DESIGN:
Intervention Model Description: Subjects are assigned to 1 of 2 or more groups in parallel for the duration of the study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): Subjects with C1-INH HAE receiving buffer only
  Interventions: Drug: Placebo
- CSL312 (low) (Active Comparator): Subjects with C1-INH HAE receiving low dose CSL312
  Interventions: Biological: Factor XIIa antagonist monoclonal antibody
- CSL312 (med) (Active Comparator): Subjects with C1-INH HAE receiving medium dose CSL312
  Interventions: Biological: Factor XIIa antagonist monoclonal antibody
- CSL312 (high) (Active Comparator): Subjects with C1-INH HAE receiving high dose CSL312
  Interventions: Biological: Factor XIIa antagonist monoclonal antibody
- CSL312 (med/high) (Active Comparator): Subjects with C1-INH HAE receiving medium/high dose CSL312
  Interventions: Biological: Factor XIIa antagonist monoclonal antibody

INTERVENTIONS:
Biological: Factor XIIa antagonist monoclonal antibody — Factor XIIa antagonist monoclonal antibody for intravenous and subcutaneous use
  Other Names: CSL312
  Arms: CSL312 (high); CSL312 (low); CSL312 (med); CSL312 (med/high)
Drug: Placebo — Buffer without active ingredient
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, placebo-controlled, parallel-arm, phase 2 study to investigate the clinical efficacy, pharmacokinetics, and safety of CSL312 as prophylaxis to prevent attacks in subjects with HAE.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged ≥ 18 to ≤ 65 years
* A diagnosis of C1-INH HAE or FXII/PLG HAE;
* For subjects with C1-INH HAE: ≥ 4 HAE attacks over a consecutive 2-month period during the 3 months before Screening, as documented in the subject's medical record.

Exclusion Criteria:

* History of clinically significant arterial or venous thrombosis, or current clinically significant prothrombotic risk
* History of an uncontrolled, abnormal bleeding event due to a coagulopathy, or a current clinically significant coagulopathy or clinically significant risks for bleeding events
* Known incurable malignancies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring LLC
Locations (16):
- United States (7):
  - Donald S. Levy, Orange, California
  - Allergy & Asthma Clinical Research, Walnut Creek, California
  - Immunoe Health Centers, Centennial, Colorado
  - Institute for Asthma and Allergy, Chevy Chase, Maryland
  - The Mount Sinai Hospital, New York, New York
  - Pennsylvania State University, Hershey, Pennsylvania
  - AARA Research Center, Dallas, Texas
- Campbelltown Hospital, Campbelltown, New South Wales, Australia
- Canada (3):
  - University of Alberta, Edmonton, Alberta
  - Allergy and Clinical Immunology McMaster University, Hamilton, Ontario
  - Ottawa Allergy Research Corp, Ottawa, Ontario
- Germany (4):
  - Charité Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Frankfurt Goethe-Universität, Frankfurt
  - Hautklinik und Poliklinik der Universitätsklinik Mainz, Mainz
  - HZRM Hämophilie Zentrum Rhein Main GmbH, Mörfelden-Walldorf
- Barzilai University Medical Center, Ashkelon, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Craig TJ, Levy DS, Reshef A, Lumry WR, Martinez-Saguer I, Jacobs JS, Yang WH, Ritchie B, Aygoren-Pursun E, Keith PK, Busse P, Feuersenger H, Alexandru Bica M, Jacobs I, Pragst I, Magerl M. Garadacimab for hereditary angioedema attack prevention: long-term efficacy, quality of life, and safety data from a phase 2, randomised, open-label extension study. Lancet Haematol. 2024 Jun;11(6):e436-e447. doi: 10.1016/S2352-3026(24)00081-4. Epub 2024 May 3. PMID 38710185
- [Derived] Beard N, Frese M, Smertina E, Mere P, Katelaris C, Mills K. Interventions for the long-term prevention of hereditary angioedema attacks. Cochrane Database Syst Rev. 2022 Nov 3;11(11):CD013403. doi: 10.1002/14651858.CD013403.pub2. PMID 36326435
- [Derived] Craig T, Magerl M, Levy DS, Reshef A, Lumry WR, Martinez-Saguer I, Jacobs JS, Yang WH, Ritchie B, Aygoren-Pursun E, Keith PK, Busse P, Feuersenger H, Pawaskar D, Jacobs I, Pragst I, Doyle MK. Prophylactic use of an anti-activated factor XII monoclonal antibody, garadacimab, for patients with C1-esterase inhibitor-deficient hereditary angioedema: a randomised, double-blind, placebo-controlled, phase 2 trial. Lancet. 2022 Mar 5;399(10328):945-955. doi: 10.1016/S0140-6736(21)02225-X. Epub 2022 Feb 24. PMID 35219377

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Treatment Period 1 participants were assigned to 1 of 5 treatment arms. Treatment period 2 participants that completed Treatment Period 1 were assigned to either CSL312 (medium) or CSL312 (high) and could be up-titrated from CSL312 (medium) to CSL312 (med/high), if necessary. They were down-titrated from CSL312 (high) to CSL312 (medium). Only 2 subjects from the CSL312 (FXII/PLG HAE) arm were treated with CSL312 in Treatment Period 2.
Groups:
- Placebo: Subjects with C1-INH HAE (Hereditary angioedema with C1-esterase inhibitor deficiency) receiving buffer only
  Placebo: Buffer without active ingredient
- CSL312 (Low): Subjects with C1-INH HAE (Hereditary angioedema with C1-esterase inhibitor deficiency) receiving low dose CSL312
  Factor XIIa antagonist monoclonal antibody: Factor XIIa antagonist monoclonal antibody for intravenous and subcutaneous use
- CSL312 (Med): Subjects with C1-INH HAE (Hereditary angioedema with C1-esterase inhibitor deficiency) receiving medium dose CSL312
  Factor XIIa antagonist monoclonal antibody: Factor XIIa antagonist monoclonal antibody for intravenous and subcutaneous use
- CSL312 (High): Subjects with C1-INH HAE (Hereditary angioedema with C1-esterase inhibitor deficiency) receiving high dose CSL312
  Factor XIIa antagonist monoclonal antibody: Factor XIIa antagonist monoclonal antibody for intravenous and subcutaneous use
- CSL312 (Med/High): Subjects with C1-INH HAE (Hereditary angioedema with C1-esterase inhibitor deficiency) receiving medium/high dose CSL312
  Factor XIIa antagonist monoclonal antibody: Factor XIIa antagonist monoclonal antibody for intravenous and subcutaneous use
- CSL312 (FXII/PLG HAE): Subjects with FXII/PLG HAE (Hereditary Angioedema with Normal C1-esterase Inhibitor and Factor XII or Plasminogen Gene Mutation) receiving high dose CSL312
Period: Treatment Period 1
Arm/Group | Placebo | CSL312 (Low) | CSL312 (Med) | CSL312 (High) | CSL312 (Med/High) | CSL312 (FXII/PLG HAE)
Started | 8 | 9 | 8 | 7 | 6 | 6
Completed | 8 | 9 | 8 | 7 | 6 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 1
Period: Treatment Period 2
Arm/Group | Placebo | CSL312 (Low) | CSL312 (Med) | CSL312 (High) | CSL312 (Med/High) | CSL312 (FXII/PLG HAE)
Started | 0 | 0 | 20 | 18 | 0 | 2
Completed | 0 | 0 | 20 | 16 | 0 | 2
Not Completed | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population consisted of all subjects who provided informed consent, underwent any study screening procedure, and who were assigned to treatment in Treatment Period 1 or to treatment in Treatment Period 2, regardless of whether they received investigational product.
Groups:
- CSL312 (Low): Subjects with C1-INH HAE (Hereditary angioedema with C1-esterase inhibitor deficiency)receiving low dose CSL312
  Factor XIIa antagonist monoclonal antibody: Factor XIIa antagonist monoclonal antibody for intravenous and subcutaneous use
- CSL312 (High): Subjects with C1-INH HAE (Hereditary angioedema with C1-esterase inhibitor deficiency)receiving high dose CSL312
  Factor XIIa antagonist monoclonal antibody: Factor XIIa antagonist monoclonal antibody for intravenous and subcutaneous use
- Total: Total of all reporting groups
Arm/Group | Placebo | CSL312 (Low) | CSL312 (Med) | CSL312 (High) | CSL312 (Med/High) | CSL312 (FXII/PLG HAE) | Total
Number analyzed (Participants) | 8 | 9 | 8 | 7 | 6 | 6 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 8 | 6 | 6 | 6 | 43
  >=65 years | 0 | 0 | 0 | 1 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 2 | 5 | 3 | 6 | 27
  Male | 4 | 2 | 6 | 2 | 3 | 0 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1 | 0 | 2
  Not Hispanic or Latino | 7 | 9 | 8 | 7 | 5 | 6 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 2 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White | 7 | 9 | 8 | 5 | 4 | 6 | 39
  More than one race | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 1 | 3 | 2 | 1 | 0 | 0 | 7
  United States | 4 | 2 | 0 | 2 | 2 | 1 | 11
  Israel | 0 | 2 | 2 | 1 | 2 | 2 | 9
  Germany | 3 | 2 | 4 | 3 | 2 | 3 | 17

OUTCOME MEASURES:

1. Primary Outcome: The Mean Time Normalized Number of HAE Attacks Per Month in Subjects With C1-INH HAE During Treatment Period 1
Description: The time-normalized number of HAE attacks per month during Treatment Period 1 for a subject was calculated as the (number of HAE attacks / length of subject's evaluation period in days) * 30.4375
Time Frame: 13 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Number of HAE attacks per month
Arm/Group | Placebo | CSL312 (Low) | CSL312 (Med) | CSL312 (High) | CSL312 (Med/High)
Number analyzed (Participants) | 8 | 9 | 8 | 7 | 6
Number of HAE attacks per month | 4.24 (1.801) | 0.48 (1.057) | 0.05 (0.127) | 0.35 (0.407) | 0.14 (0.222)

2. Secondary Outcome: The Number of Responder Subjects With C1-INH HAE During Treatment Period 1
Description: Response is defined as a ≥ 50% relative reduction in the time-normalized number of HAE attacks (per month) during Treatment Period 1 compared to each subject's time-normalized number of HAE attacks (per month) during the Run-in Period
Time Frame: 13 weeks
Population: ITT
Measure: Number; unit: Number of participants
Arm/Group | Placebo | CSL312 (Low) | CSL312 (Med) | CSL312 (High) | CSL312 (Med/High)
Number analyzed (Participants) | 8 | 9 | 8 | 7 | 6
Number of participants | 0 | 9 | 8 | 6 | 6

3. Secondary Outcome: The Percentage of Responder Subjects With C1-INH HAE During Treatment Period 1
Description: as for outcome 2
Time Frame: 13 weeks
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | CSL312 (Low) | CSL312 (Med) | CSL312 (High) | CSL312 (Med/High)
Number analyzed (Participants) | 8 | 9 | 8 | 7 | 6
percentage of participants | 0 | 100.0 | 100.0 | 85.7 | 100.0

4. Secondary Outcome: The Number of HAE Attack-free Subjects With C1-INH HAE During Treatment Period 1
Time Frame: 13 weeks
Population: ITT
Measure: Number; unit: Number of participants
Arm/Group | Placebo | CSL312 (Low) | CSL312 (Med) | CSL312 (High) | CSL312 (Med/High)
Number analyzed (Participants) | 8 | 9 | 8 | 7 | 6
Number of participants | 0 | 5 | 7 | 3 | 4

5. Secondary Outcome: The Percentage of HAE Attack-free Subjects With C1-INH HAE During Treatment Period 1
Time Frame: 13 weeks
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | CSL312 (Low) | CSL312 (Med) | CSL312 (High) | CSL312 (Med/High)
Number analyzed (Participants) | 8 | 9 | 8 | 7 | 6
percentage of participants | 0 | 55.6 | 87.5 | 42.9 | 66.7

6. Secondary Outcome: The Number of Mild, Moderate or Severe HAE Attacks in Subjects With C1-INH HAE During Treatment Period 1
Time Frame: 13 weeks
Population: ITT
Measure: Number; unit: Number of HAE attacks
Units Other Than Participants: Total Number of HAE Attacks
Arm/Group | Placebo | CSL312 (Low) | CSL312 (Med) | CSL312 (High) | CSL312 (Med/High)
Number analyzed (Participants) | 8 | 9 | 8 | 7 | 6
Number analyzed (Total Number of HAE Attacks) | 95 | 12 | 1 | 7 | 2
Number of HAE attacks
  Mild | 32 | 3 | 0 | 2 | 2
  Moderate | 43 | 9 | 1 | 4 | 0
  Severe | 20 | 0 | 0 | 1 | 0

7. Secondary Outcome: The Percentage of Mild, Moderate or Severe HAE Attacks in Subjects With C1-INH HAE During Treatment Period 1
Time Frame: 13 weeks
Population: ITT
Measure: Number; unit: percentage of HAE attacks
Units Other Than Participants: Total Number of HAE Attacks
Arm/Group | Placebo | CSL312 (Low) | CSL312 (Med) | CSL312 (High) | CSL312 (Med/High)
Number analyzed (Participants) | 8 | 9 | 8 | 7 | 6
Number analyzed (Total Number of HAE Attacks) | 95 | 12 | 1 | 7 | 2
percentage of HAE attacks
  Mild | 33.7 | 25.0 | 0 | 28.6 | 100.0
  Moderate | 45.3 | 75.0 | 100.0 | 57.1 | 0
  Severe | 21.1 | 0 | 0 | 14.3 | 0

8. Secondary Outcome: The Mean Time-normalized Number of Mild, Moderate or Severe HAE Attacks Per Month in Subjects With C1-INH HAE During Treatment Period 1
Description: as for outcome 1
Time Frame: 13 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: Number of HAE attacks per month
Units Other Than Participants: Total number of HAE attacks
Arm/Group | Placebo | CSL312 (Low) | CSL312 (Med) | CSL312 (High) | CSL312 (Med/High)
Number analyzed (Participants) | 8 | 9 | 8 | 7 | 6
Number analyzed (Total number of HAE attacks) | 95 | 12 | 1 | 7 | 2
Number of HAE attacks per month
  Mild | 1.42 (1.395) | 0.12 (0.177) | 0.0 (0.000) | 0.10 (0.168) | 0.14 (0.222)
  Moderate | 1.93 (1.403) | 0.36 (1.087) | 0.05 (0.127) | 0.20 (0.347) | 0.0 (0.000)
  Severe | 0.89 (1.365) | 0.0 (0.000) | 0.0 (0.000) | 0.05 (0.136) | 0.0 (0.000)

9. Secondary Outcome: The Number of Subjects With at Least One (1) HAE Attack Treated With On-demand HAE Medication, in Subjects With C1-INH HAE During Treatment Period 1
Time Frame: 13 weeks
Population: ITT
Measure: Number; unit: Number of participants
Arm/Group | Placebo | CSL312 (Low) | CSL312 (Med) | CSL312 (High) | CSL312 (Med/High)
Number analyzed (Participants) | 8 | 9 | 8 | 7 | 6
Number of participants | 8 | 3 | 1 | 2 | 0

10. Secondary Outcome: The Percentage of Subjects With at Least One (1) HAE Attack Treated With On-demand HAE Medication, in Subjects With C1-INH HAE During Treatment Period 1
Time Frame: 13 weeks
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | CSL312 (Low) | CSL312 (Med) | CSL312 (High) | CSL312 (Med/High)
Number analyzed (Participants) | 8 | 9 | 8 | 7 | 6
percentage of participants | 100.0 | 33.3 | 12.5 | 28.6 | 0

11. Secondary Outcome: Maximum Concentration (Cmax) of CSL312 in Subjects With C1-INH HAE During Treatment Period 1
Time Frame: 13 weeks
Population: The pharmacokinetic (PK) population consisted of all subjects in the Safety population for whom at least 1 measurable concentration of CSL312 was reported.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Placebo | CSL312 (Low) | CSL312 (Med) | CSL312 (High) | CSL312 (Med/High)
Number analyzed (Participants) | 0 | 9 | 8 | 7 | 0
ug/mL |  | 10.6 (6.09) | 15.9 (5.22) | 56.4 (15.9) |

12. Secondary Outcome: Area Under the Concentration-time Curve in 1 Dosing Interval (AUC0-tau) of CSL312 in Subjects With C1-INH HAE During Treatment Period 1
Time Frame: 13 weeks
Population: PK
Measure: Mean (Standard Deviation); unit: h*μg/mL
Arm/Group | Placebo | CSL312 (Low) | CSL312 (Med) | CSL312 (High) | CSL312 (Med/High)
Number analyzed (Participants) | 0 | 9 | 8 | 7 | 0
h*μg/mL |  | 4507 (2424) | 7166 (2410) | 26514 (8151) |

13. Secondary Outcome: Time of Maximum Concentration (Tmax) of CSL312 in Subjects With C1-INH HAE During Treatment Period 1
Time Frame: 13 weeks
Population: PK
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo | CSL312 (Low) | CSL312 (Med) | CSL312 (High) | CSL312 (Med/High)
Number analyzed (Participants) | 0 | 9 | 8 | 7 | 0
hours |  | 143.38 [45.4 to 196] | 165.51 [116 to 218] | 165.63 [72.4 to 188] |

14. Secondary Outcome: Terminal Elimination Half-life (T1/2) of CSL312 in Subjects With C1-INH HAE During Treatment Period 1
Time Frame: 13 weeks
Population: PK
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Placebo | CSL312 (Low) | CSL312 (Med) | CSL312 (High) | CSL312 (Med/High)
Number analyzed (Participants) | 0 | 7 | 7 | 5 | 0
hours |  | 411.7 (96.97) | 394.0 (85.64) | 443.5 (44.00) |

15. Secondary Outcome: Clearance (CL/F) of CSL312 in Subjects With C1-INH HAE During Treatment Period 1
Time Frame: 13 weeks
Population: PK
Measure: Mean (Standard Deviation); unit: L/hour
Arm/Group | Placebo | CSL312 (Low) | CSL312 (Med) | CSL312 (High) | CSL312 (Med/High)
Number analyzed (Participants) | 0 | 9 | 8 | 7 | 0
L/hour |  | 0.0198 (0.0079) | 0.0303 (0.0084) | 0.0246 (0.0079) |

16. Secondary Outcome: Volume of Distribution During the Elimination Phase (Vz/F) of CSL312 in Subjects With C1-INH HAE During Treatment Period 1
Time Frame: 13 weeks
Population: PK
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Placebo | CSL312 (Low) | CSL312 (Med) | CSL312 (High) | CSL312 (Med/High)
Number analyzed (Participants) | 0 | 7 | 7 | 5 | 0
Liters |  | 10.6 (5.10) | 17.0 (4.78) | 17.1 (6.67) |

17. Secondary Outcome: The Number of Subjects With C1-INH HAE With Adverse Events (AEs), Serious Adverse Events (SAEs), Adverse Events of Special Interest (AESI), Injection Site Reactions (ISRs), Binding Antibodies to CSL312 During Treatment Period 1
Description: Adverse events of special interest is defined as anaphylaxis, thromboembolic events, and bleeding events.
Time Frame: 13 weeks
Population: The Safety population (SP) consisted of all subjects who provided informed consent, were assigned to treatment in Treatment Period 1 or to treatment in Treatment Period 2 and received at least 1 dose or partial dose of investigational product and was based on the actual treatment received.
Measure: Number; unit: Number of participants
Arm/Group | Placebo | CSL312 (Low) | CSL312 (Med) | CSL312 (High) | CSL312 (Med/High)
Number analyzed (Participants) | 8 | 9 | 8 | 7 | 6
Number of participants
  AEs | 7 | 7 | 7 | 7 | 4
  SAEs | 0 | 0 | 0 | 0 | 0
  AESI | 1 | 0 | 0 | 0 | 0
  ISRs | 2 | 1 | 1 | 4 | 2
  Binding Antibodies to CSL312 | 1 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Approximately 129 weeks per participant
Description: Adverse events were collected for both Treatment Periods 1 (up to 13 weeks) and 2 (up to 44 weeks + up to 13 weeks follow-up). Adverse events will be reported by Treatment Period.
Groups:
- CSL312 (Med-Period 2): Subjects with C1-INH HAE receiving medium dose CSL312
- CSL312 (Med/High-Period 2): Subjects with C1-INH HAE receiving medium/high dose CSL312
- CSL312 (High-Period 2): Subjects with C1-INH HAE receiving high dose CSL312
- CSL312 (FXII/PLG HAE-Period 1); CSL312 (FXII/PLG HAE-Period 2): Subjects with FXII/PLG HAE (Hereditary Angioedema with Normal C1-esterase Inhibitor and Factor XII or Plasminogen Gene Mutation) receiving high dose CSL312
Arm/Group | Placebo | CSL312 (Low) | CSL312 (Med) | CSL312 (High) | CSL312 (Med/High) | CSL312 (Med-Period 2) | CSL312 (Med/High-Period 2) | CSL312 (High-Period 2) | CSL312 (FXII/PLG HAE-Period 1) | CSL312 (FXII/PLG HAE-Period 2)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9 | 0/8 | 0/7 | 0/6 | 0/36 | 0/3 | 0/18 | 0/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9 | 0/8 | 0/7 | 0/6 | 1/36 | 0/3 | 1/18 | 1/6 | 0/2
Other Adverse Events (participants affected / at risk) | 7/8 | 7/9 | 7/8 | 7/7 | 4/6 | 25/36 | 2/3 | 17/18 | 1/6 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | CSL312 (Low) (N=9) | CSL312 (Med) (N=8) | CSL312 (High) (N=7) | CSL312 (Med/High) (N=6) | CSL312 (Med-Period 2) (N=36) | CSL312 (Med/High-Period 2) (N=3) | CSL312 (High-Period 2) (N=18) | CSL312 (FXII/PLG HAE-Period 1) (N=6) | CSL312 (FXII/PLG HAE-Period 2) (N=2)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hereditary angioedema (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | CSL312 (Low) (N=9) | CSL312 (Med) (N=8) | CSL312 (High) (N=7) | CSL312 (Med/High) (N=6) | CSL312 (Med-Period 2) (N=36) | CSL312 (Med/High-Period 2) (N=3) | CSL312 (High-Period 2) (N=18) | CSL312 (FXII/PLG HAE-Period 1) (N=6) | CSL312 (FXII/PLG HAE-Period 2) (N=2)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 3 (6) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (6) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (4) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site urticaria (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polymorphic light eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 2 (5) | 6 (12) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Anosmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plantar fascial fibromatosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular access site bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Initial insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pregnancy of partner (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-03-20): https://cdn.clinicaltrials.gov/large-docs/28/NCT03712228/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-19): https://cdn.clinicaltrials.gov/large-docs/28/NCT03712228/SAP_001.pdf